CLINICAL TRIAL: NCT07266077
Title: Influence Of A Slope Adaptive Foot On Participation Of Veterans With Lower-Limb Amputations
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: RRD4-004-24W
Record Dates: First submitted 2025-11-20; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Amputation
Keywords: Artificial Limbs; Amputation; Leg Prosthesis; Ankle; Community Participation; Social Participation; Falls

STUDY DESIGN:
Intervention Model Description: This study includes two distinct phases. The first is a cross-over randomized controlled trial (RCT) with a four-week take-home period to test two hydraulic foot types: the SAF and a typical hydraulic foot (Fillauer Motion Foot SLX). The second phase of this study is a one-year observational period of the Veteran's preferred foot (ESAR, SAF, or SLX).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SAF-SLX (Experimental): Participants in this arm will start the cross-over randomized controlled trial with the SAF. After a four-week take-home period with the SAF, participants will return to their usual prosthetic foot for a four-week washout period. They will then be fit with the SLX for a four-week take-home period.
  Interventions: Device: Fillauer Slope Adaptive Foot; Device: Fillauer Motion Foot SLX
- SLX-SAF (Experimental): Participants in this arm will start the cross-over randomized controlled trial with the SLX. After a four-week take-home period with the SLX, participants will return to their usual prosthetic foot for a four-week washout period. They will then be fit with the SAF for a four-week take-home period.
  Interventions: Device: Fillauer Slope Adaptive Foot; Device: Fillauer Motion Foot SLX

INTERVENTIONS:
Device: Fillauer Slope Adaptive Foot — The SAF uses an articulated ankle and damped plantarflexion to accommodate slopes and uneven terrain. It locks when the forefoot reaches the ground at the beginning of stance phase, which allows the SAF to re-align, or adapt, to the walking surface. After the SAF locks, the laminated foot plate can deflect and store energy as dorsiflexion occurs, returning that energy to the user in late stance for forward propulsion. Finally, at the end of stance phase, when the toe leaves the ground, the SAF unlocks and actively dorsiflexes the ankle to increase toe clearance during swing.
  Other Names: SAF
Device: Fillauer Motion Foot SLX — The SLX is an articulated, hydraulic ankle that provides passive ankle motion through damped plantarflexion and dorsiflexion to facilitate slope accommodation.
  Other Names: SLX

SUMMARY:
Veterans with below-knee amputations are limited by prosthetic feet that cannot adapt to sloped and uneven terrain. This limitation results in reduced mobility, reduced balance confidence, and a higher risk of falls among some individuals who use below-knee prostheses, which have been shown to negatively impact participation in daily and recreational activities. The investigative group has designed a novel Slope Adaptive Foot (SAF) that is mechanically passive, capable of slope adaption on every step of walking, and maintains high levels of energy storage and return. Pilot testing of the SAF with Veterans has generated excellent results to date, with comments suggesting potential improvements in participation. This study will evaluate the extent to which participation and fall-related health outcomes are influenced by using the SAF versus a typical hydraulic foot in a cross-over randomized controlled trial. Using mixed-methods, the investigators will also collect long-term data of Veterans using their preferred foot to inform the development of evidence-based education materials for use in clinical decision making.

DETAILED DESCRIPTION:
Background and Relevance to VA - Over 90% of Veterans who use a below-knee prosthesis in the community are prescribed an energy storage and return (ESAR) foot. ESAR feet are designed to assist with forward propulsion during walking, which many users find helpful for certain activities. However, ESAR feet lack ankle articulation, making it difficult to walk on non-level surfaces. To overcome this limitation, typical hydraulic feet incorporate damped ankle motion to accommodate walking on uneven terrain. While potentially improving aspects of participation and fall-related health, typical hydraulic feet have reduced energy storage and return compared to ESAR feet.

To combine the benefits of ESAR and typical hydraulic feet, the Minneapolis VA, in collaboration with Fillauer Motion Control, Inc., has developed a novel hydraulic Slope Adaptive Foot (SAF). During pilot testing, most Veterans preferred the SAF over their prescribed ESAR foot and reported improvements in participation. Further research is needed to evaluate the impact of different prosthetic feet on participation and fall-related health in order to identify which patients are best suited for an ESAR foot, a typical hydraulic foot, or the SAF.

Innovation and Impact - The long-term goal of this project is to inform prescription of hydraulic feet for Veterans living with lower-limb amputation to optimize their participation in important life roles and activities. Results of this study will help to develop evidence-based provider training and patient education materials to assist with precision rehabilitation and a patient-centered care approach to prescribing hydraulic prosthetic feet.

Aim 1 - Evaluate the influence of different prosthetic foot-related factors on participation. PROMIS Ability to Participate in Social Roles and Activities (APSRA) and PROMIS Satisfaction with Social Roles and Activities (SSRA) will be administered during a cross-over randomized control trial (RCT). This aim will test the hypothesis that using the SAF will be associated with greater PROMIS-APSRA and/or PROMIS-SSRA scores relative to a typical hydraulic foot and that using either hydraulic foot will be associated with greater PROMIS-APSRA and/or PROMIS-SSRA scores compared to the ESAR foot.

Aim 2 - Characterize the lived experiences of Veterans using their preferred prosthetic foot to inform clinical decision making. Mixed-methods will be used to explore how participation in social roles and activities is influenced by hydraulic and ESAR feet. Gaining a deeper understanding of Veterans' experiences across a range of situations and environments will inform the development of evidence-based education materials.

Exploratory Aim - Evaluate the influence of different prosthetic foot-related factors on fall-related health outcomes. The Prosthetic Limb Users Survey of Fall-Related Health (PLUS-FRH), which includes four distinct and important domains, will be administered during a cross-over RCT. This aim will test the hypothesis that using the SAF will be associated with improved fall-related health outcomes relative to a typical hydraulic foot and that using either hydraulic foot will be associated with improved fall-related health outcomes compared to the ESAR foot.

Methodology - To address these aims, this study will 1) conduct a cross-over RCT of the SAF versus a typical hydraulic foot (Motion Foot SLX, Fillauer) among 30 Veterans with a below-knee amputation who use an ESAR foot and have no prior experience with a hydraulic foot, and 2) conduct a one-year observational study in which Veterans use their preferred prosthetic foot. Participants will complete quantitative (PROMIS-APSRA, PROMIS-SSRA, PLUS-FRH) and qualitative (semi-structured interviews) assessments at baseline and after each period of the cross-over RCT and quarterly during the one-year observational study. A participatory method will be used in which Veterans will be asked to share photos with a short narrative to portray their experiences with their preferred prosthetic foot to prompt discussion during the quarterly interviews of the one-year observational study.

Participating Sites - Minneapolis VA Health Care System (data collection site) and the University of Washington.

Duration of Participant Intake (Study Duration) - This project is projected to occur over four years. The project will begin with a 3-month start-up period and recruitment will continue for 18 months following start-up. Data collection will conclude with 9 months remaining in the study timeline, which will be used for data analysis, dissemination, development of implementation materials, and study closure.

Path to Implementation - Data gathered from this study will be used to draft evidence-based education materials for providers and Veterans. These materials, which will provide pertinent and useful information about foot options (ESAR, SLX, SAF) for prosthetic prescription, will be used in a future implementation study.

ELIGIBILITY:
Inclusion Criteria:

* US military Veterans willing to travel to the Minneapolis VA Health Care System
* Unilateral, below-knee amputation
* Use of a definitive prosthesis for at least 12 months (limb volume has stabilized and has accommodated to prosthesis use post-amputation)
* Medicare Functional Classification Level K3 ambulator (unlimited community ambulator)
* Well-fitting and well-aligned prosthesis
* Uses a prescribed energy storage and return foot (ESAR)
* Blessed Orientation-Memory-Concentration (Short Blessed) test score between 0-6 (no cognitive impairment)
* Access to computer, tablet, or smartphone and internet for video conferencing and REDCap data collection

Exclusion Criteria:

* Residual-limb skin problems
* Not a regular prosthesis user
* Mass over 125 kg (275 lbs)
* Residual limb too long to accommodate the study feet (104 mm of build height)
* Has used a hydraulic foot previously as part of clinical care or a research study
* Documented major neurocognitive disorder (i.e., dementia) with evidence of impact on activities of daily living and/or instrumental activities of daily living
* Baseline PROMIS-APSRA or PROMIS-SSRA scores at the maximum levels (no room for improvement on primary outcomes)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
PROMIS Ability to Participate in Social Roles and Activities (APSRA) | Day 1 of the RCT, after each 4-week intervention in the RCT, and 13 weeks, 26 weeks, 39 weeks, and 52 weeks into the 1-year observational period of the study
  This Patient Reported Outcome Measurement Information System (PROMIS) short form is an 8-item self-report survey instrument, developed from PROMIS item banks, that provides T scores (mean = 50, SD = 10) based on a normative sample from a general population of healthy US adults. The PROMIS-APSRA specifically measures the frequency with which one has trouble with completing or needs to limit participation in social roles and activities, including leisure activities and activities with friends and family. This PROMIS measure uses a 5-point ordinal response scale, where higher values indicate a higher degree of ability to participate.
PROMIS Satisfaction with Social Roles and Activities (SSRA) | Day 1 of the RCT, after each 4-week intervention in the RCT, and 13 weeks, 26 weeks, 39 weeks, and 52 weeks into the 1-year observational period of the study
  This Patient Reported Outcome Measurement Information System (PROMIS) short form is an 8-item self-report survey instrument, developed from PROMIS item banks, that provides T scores (mean = 50, SD = 10) based on a normative sample from a general population of healthy US adults. The PROMIS-SSRA measures the level of satisfaction with one's ability to participate in recreational activities, activities of daily living, and to meet the needs of friends and family. This PROMIS measure uses a 5-point ordinal response scale, where higher values indicate a higher degree of satisfaction with participation.

SECONDARY OUTCOMES:
Prosthetic Limb Users Survey of Fall-Related Health (PLUS-FRH) | Day 1 of the RCT, after each 4-week intervention in the RCT, and 13 weeks, 26 weeks, 39 weeks, and 52 weeks into the 1-year observational period of the study
  Each domain of the PLUS-FRH (fall-related self-efficacy, anxiety, avoidance behavior, and interference) corresponds to a 15-item instrument that provides T scores (mean = 50, SD = 10) based on a normative sample of lower-limb prosthesis users. The items on the PLUS-FRH use a 5-point ordinal response scale, where higher values correspond to better or worse fall-related health outcomes, depending on the domain.

OTHER OUTCOMES:
Timed Up and Go (TUG) | Day 1 of the RCT, after each 4-week intervention in the RCT, and at the end of the 1-year observational period of the study
  The TUG is test protocol for balance function. From a seated position in a standard armchair, the participant is asked to do the following: 1) stand up from the chair, 2) walk to a line on the floor 10 feet away at a normal pace, 3) turn, 4) walk back to the chair at a normal pace, 5) sit down again. Performance is measured as the time it takes to complete the test.
10-meter Walk Test (10MWT) | Day 1 of the RCT, after each 4-week intervention in the RCT, and at the end of the 1-year observational period of the study
  Gait speed (10-meter walk using the middle 6 meters) is assessed under two conditions: 1) normal speed and 2) fastest speed. A difference of 0.10 m/s is defined as the minimal clinically important difference.
Modified Five-Time Sit-to-Stand (m5xSTS) | Day 1 of the RCT, after each 4-week intervention in the RCT, and at the end of the 1-year observational period of the study
  The m5xSTS test assesses functional lower extremity strength and transitional movements. The participant is instructed to sit with arms resting on their lap and back against a chair. They are instructed to stand up and sit down five times as quickly as possible when prompted. The time taken to complete the test is recorded. If needed, the participant can use armrests or a walker, the use of which should be documented.
Prosthetic Limb Users Survey of Mobility (PLUS-M) | Day 1 of the RCT, after each 4-week intervention in the RCT, and at the end of the 1-year observational period of the study
  The PLUS-M is a 12-item instrument that measures prosthesis users' mobility (i.e., their ability to move intentionally and independently from one place to another). Individual PLUS-M questions assess respondents' perceived ability to carry out specific activities that require use of both lower limbs. PLUS-M questions cover movements that range from basic ambulation (e.g., walking a short distance indoors) to complex activities (e.g., hiking for long distances over uneven ground). The items on the PLUS-M use a 5-point ordinal response scale that reflects the degree of difficulty with which respondents report they can carry out these activities. PLUS-M T scores (mean = 50, SD = 10) are based on a normative sample of lower-limb prosthesis users.
Prosthetic Limb Users Survey of Mobility-Terrain (PLUS-M Terrain) | Day 1 of the RCT, after each 4-week intervention in the RCT, and at the end of the 1-year observational period of the study
  The PLUS-M Terrain is an 18-item instrument that measures prosthesis users' mobility (i.e., their ability to move intentionally and independently from one place to another) on different terrain. Individual PLUS-M Terrain questions assess respondents' perceived ability to carry out specific activities that require use of both lower limbs. PLUS-M Terrain questions cover movements that range from basic ambulation (e.g., walking across a parking lot) to complex activities (e.g., hiking steep mountainous terrain). The items on the PLUS-M Terrain use a 5-point ordinal response scale that reflects the degree of difficulty with which respondents report they can carry out these activities. PLUS-M T scores (mean = 50, SD = 10) are based on a normative sample of lower-limb prosthesis users.
Socket Comfort Score (SCS) | Day 1 of the RCT, after each 4-week intervention in the RCT, and 13 weeks, 26 weeks, 39 weeks, and 52 weeks into the 1-year observational period of the study
  The SCS is a subjective measure where respondents report their comfort level with a prosthetic socket. The score ranges from 0 (most uncomfortable) to 10 (most comfortable).
WHODAS 2.0-Modified | Day 1 of the RCT, after each 4-week intervention in the RCT, and 13 weeks, 26 weeks, 39 weeks, and 52 weeks into the 1-year observational period of the study
  The WHODAS 2.0 asks respondents about difficulties due to health/mental health conditions. The modified version covers 5 domains of functioning: mobility, self-care, getting along, life activities, and participation. The items on the WHODAS 2.0 use a 5-point ordinal response scale and two scoring methods can be used: 1) score (and its percentile) and 2) average score (and its descriptor).
Activities-Specific Balance Confidence (ABC) | Day 1 of the RCT, after each 4-week intervention in the RCT, and at the end of the 1-year observational period of the study
  The ABC scale is a self-report measure used to assess an individual's confidence in performing various activities without losing balance or experiencing unsteadiness. In consists for 16 activities, ranging from common tasks like walking around the house to more challenging situations such as stepping off a moving escalator while carrying packages. Items are rated on a rating scale that ranges from 0 to 100. The overall score is calculated by adding item scores, then dividing by the total number of items.
Amputee Body Image Scale-Revised (ABIS-R) | Day 1 of the RCT, after each 4-week intervention in the RCT, and at the end of the 1-year observational period of the study
  The ABIS-R was developed to measure body image perceptions in individuals who have undergone amputations. It consists of 14 items that evaluate various aspects of body image, including feelings of self-esteem, anxiety, and overall psychosocial well-being related to changes in body image after limb loss. The ABIS-R uses a three-level response scale scored from 1 (none of the time) to 5 (all of the time), with total scores ranging from 14 to 70 where higher scores indicate greater body image disturbance.
PROMIS Pain Interference 8a | Day 1 of the RCT, after each 4-week intervention in the RCT, and at the end of the 1-year observational period of the study
  The PROMIS Pain Interference 8a is a validated self-report tool to assess how pain impacts an individual's daily activities and enjoyment of life. It consists of 8 items that ask respondents to rate how much pain has interfered with life activities over the past 7 days using a 5-point scale (1=not at all, 5= very much). The raw scores are converted to T scores with higher scores indicating greater pain interference.
PROMIS Depression 8a | Day 1 of the RCT, after each 4-week intervention in the RCT, and at the end of the 1-year observational period of the study
  The PROMIS Depression 8a is a validated self-report tool to assess depressive symptoms in individuals aged 18 and older. It consists of 8 items that ask respondents to rate the severity of their depression symptoms over the past 7 days using a 5-point scale (1=never, 5=always). The raw scores are converted to T scores with higher scores indicating greater severity of depression.
Prosthetic Foot Preference Rating Scales | Day 1 of the RCT and after each 4-week intervention in the RCT
  The Prosthetic Foot Preference Rating Scales are designed to evaluate the experiential preference of users for different prosthetic feet. The tool includes 9 distinct numeric rating scales to assess users' prosthetic foot preferences after trials of different feet. Six of the scales are activity-specific rating scales intended to measure users' perceived ability to perform a specific activity. Three global scales are intended to evaluate more holistic aspects of users' experience. All scales use an 11-point numeric rating (0-10) that include descriptive anchors at 0 and 10 to characterize the extreme ends of the scale. Scores from the activity-specific scales can be averaged into a mean activity rating score, whereas scores from the global scale are not intended to be combined into a summary score.
Self-Administered Comorbidity Questionnaire (SCQ) | Day 1 of the RCT and Day 1, 26 weeks, and 52 weeks into the 1-year observational period of the study
  The SCQ consists of a series of questions regarding common health problems. Respondents indicate whether they currently have these problems, if they receive treatment for them, and whether these conditions limit their activities. The questionnaire addresses various body systems and includes conditions such as heart disease, high blood pressure, lung disease, and diabetes, among others.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Koehler-McNicholas, PhD MS BS, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN; Mary E Matsumoto, MD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No